CLINICAL TRIAL: NCT01178658
Title: Busulfan, Etoposide, Cytarabine, and Melphalan (BuEAM) as a Conditioning for Autologous Stem Cell Transplantation in Patients With T Cell or NK Cell Lymphoma
Brief Title: Study of Busulfan, Etoposide, Cytarabine, and Melphalan (BuEAM) Conditioning for Autologous Stem Cell Transplantation (ASCT) to Treat T Cell or Natural Killer (NK) Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Inje University (Other); Severance Hospital (Other); Asan Medical Center (Other); Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Sung-Soo Yoon, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BuEAM-NK/T
Record Dates: First submitted 2010-08-03; First posted 2010-08-10 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Busulfan; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BuEAM (Experimental): Busulfan 3.2 mg/kg/d for 2 days, etoposide 400 mg/m2/d for 2 days, cytarabine 1 g/m2 for 2 days, and melphalan 140 mg/m2 for 1 day
  Interventions: Drug: Busulfan, etoposide, cytarabine, and melphalan

INTERVENTIONS:
Drug: Busulfan, etoposide, cytarabine, and melphalan — Busulfan 3.2 mg/kg/d for 2 days, etoposide 400 mg/m2/d for 2 days, cytarabine 1 g/m2 for 2 days, and melphalan 140 mg/m2 for 1 day

SUMMARY:
The purpose of this study is to evaluate the efficacy and toxicity of busulfan, etoposide, cytarabine and melphalan (BuEAM) as a conditioning for autologous stem cell transplantation in patients with non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
High-dose conditioning regimens commonly used in patients with non-Hodgkin lymphoma are BEAM (BCNU, etoposide, cytarabine, and melphalan), BEAC (BCNU, etoposide, cytarabine, and cyclophosphamide), CBV (cyclophosphamide, carmustine, and etoposide), and combination regimen with total body irradiation. Three-year progression free survival of patients with non-Hodgkin lymphoma received above high-dose chemotherapy followed by autologous stem cell rescue was reported as 40-50%, which is still unsatisfactory.

Busulfan (Bu)-based preparative regimens, which are commonly used with allogeneic stem cell transplantation have also been studied with autologous stem cell transplantation for lymphomas.

The development of intravenous busulfan achieved 100% bioavailability bypassing the oral route and increased safety and reliability of generating therapeutic busulfan levels, maximizing efficacy.

Recently, one prospective study showed that a combination conditioning regimen of intravenous busulfan, cyclophosphamide, and etoposide was found to be well tolerated and seemed to be effective in patients with aggressive non-Hodgkin lymphoma. Another prospective study for patients with multiple myeloma showed that intravenous busulfan plus melphalan conditioning regimen made no grade 3-4 non-hematologic complication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a high-intermediate/high risk international prognostic index at a diagnosis or with salvage chemotherapy-sensitive relapse/refractory non-Hodgkin lymphoma
* Patients with histologically confirmed T cell or NK cell lymphoma at diagnosis
* Patients who have not received therapy with high-dose chemotherapy and stem cell transplantation
* Life expectation of at least 3 months
* ECOG performance status ≤ 2
* Adequate hepatic function (serum bilirubin less than 2.0 mg/dL, AST and ALT less than three times the upper normal limit)
* Adequate renal function (serum creatinine less than 2.0 mg/dL).
* Adequate cardiac function (ejection fraction ≥ 45% on MUGA scan or echocardiogram).
* Adequate bone marrow function (ANC ≥ 1,000/mm3 and platelet count ≥ 75,000/mm3).
* All patients are fully informed about the nature and purpose of this study and informed consent should be given before the start of treatment. All patients should fully understand the right of trial abandon without any disadvantage

Exclusion Criteria:

* Patients with central nervous system involvement of lymphoma
* Patients positive for human immunodeficiency virus
* Pregnant or breast feeding woman
* Young woman without pregnancy test prior to treatment or pregnancy test reveals positive.
* Young woman without a reliable and proper contraceptive method
* Man being not willing to contraception
* Concurrent history of neoplasm other than non-Hodgkin lymphoma with life expectancy less than 3 months (except for curatively treated non-melanoma skin cancer or in-situ uterine cervix cancer).
* History of clinically significant cardiac dysfunction (e.g. congestive heart failure, symptomatic coronary artery disease, medically uncontrolled arrhythmia) or myocardial infarction within 12 months
* A psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible.
* Significant infection or uncontrolled bleeding
* Enrollment of other clinical trials within 4 weeks prior to treatment
* Any preexisting medical condition of sufficient severity to prevent full compliance with the study
* Patient being not willing to or unable to obey study protocol

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | After 3 years

SECONDARY OUTCOMES:
Overall survival | After 3 years
Response rate according to the International Working Group criteria | After 2 months
Adverse events | From start of conditioning to discharge
Pharmacogenetic study | After 3 years
  Pharmacogenetic study for predictive or prognostic markers using blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Soo Yoon, Principal Investigator — Seoul National University Hospital
Locations (5):
- South Korea (5):
  - Inje University Busan Paik Hospital, Inje University College of Medicine, Busan
  - Seoul National University Hospital, Seoul National University College of Medicine, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Seoul
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul
  - Ulsan University Hospital, University of Ulsan College of Medicine, Ulsan